CLINICAL TRIAL: NCT06448520
Title: Reference Values for the Muscle Power Sprint Test in Children Aged 5-12 Years
Brief Title: Reference Values for the Muscle Power Sprint Test
Acronym: Ref MPST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Louis Dossche, MD, PhD Candidate, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL86724.000.24; 12322 (Other: PaNaMa)
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Development, Child; Activity, Motor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle Power Sprint Test (MPST) (Experimental): All patients in this arm will be assessed through the MPST. We calculate the mean Power developed during the six short distance sprints, using time needed for each sprint and the weight of the study subject.
  Interventions: Other: Muscle Power Sprint Test

INTERVENTIONS:
Other: Muscle Power Sprint Test — The Muscle Power Sprint Test (MPST) is an easy-to-perform field test of anaerobic capacity for children and adolescents. The only necessities for the administration of this test are an open space, a stopwatch and two cones or lines. Test subjects are encouraged to perform six 15-meter sprints at a maximal pace between the two cones/lines, with a 10-second rest in between each effort. The distance covered during these short runs corresponds well to the distances children cover during daily play activities. The power that is generated with each sprint can be calculated using the formula: power = (total mass x 15 m²)/time³.

SUMMARY:
The goal of this prospective, cross-sectional study is to develop updated reference values for the Muscle Power Sprint Test (MPST) in children aged 5-12 years.

The main question it aims to answer is:

• What are reference ('normal') values for the MPST in children aged 5-12 years?

Participants will be asked to perform six short sprints of fifteen meters each, with a ten-second rest between each effort.

DETAILED DESCRIPTION:
SUMMARY Rationale: Children with congenital abnormalities face risks of below-average lung function and exercise tolerance (1-3). As the standard of care, our tertiary hospital enrolls these children in a prospective, longitudinal follow-up program from birth (4). This program involves regular assessments of overall health and development, including spirometry and exercise tolerance tests conducted by pediatric physiotherapists. Historically, the Bruce treadmill protocol was employed for testing maximal exercise tolerance in children aged 4 and above, but it presented limitations such as high muscular demands of the steep inclines and large workload increments, impacting reliability and potentially causing premature discontinuation (5).

In response, the Bruce protocol was replaced in newer follow-up program versions by the Muscle Power Sprint Test (MPST). Unlike the Bruce protocol, which assesses aerobic capacity, the MPST focuses on anaerobic exercise capacity, which is crucial for children's daily activities like playing with peers (6). Performing the MPST involves six short runs of 15 meters, from which the calculated 'mean power' serves as the primary outcome. The distance covered during these runs corresponds well to the distances children cover during daily play activities.

While Dutch norm values for children aged 6-18 exist, gathered mainly in rural areas between 2012 and 2016, the study highlights the need for updated reference values. Lifestyle changes, exacerbated by the Covid-19 pandemic, underscore the urgency of updating exercise tolerance reference values (7). Notably, there is a current lack of established reference values for 5-year-olds undergoing MPST testing in our longitudinal follow-up program, emphasizing the need for comparative data in this age group.

Objective: Our primary goal is to establish reference values for the MPST for primary school children aged 5-12 belonging to a diverse population living in the Netherlands.

Study design: The study adopts a prospective cross-sectional design.

Study population: Primary school or after-school childcare children aged 5-12 years.

Intervention (if applicable): The MPST, which involves six 15-meter sprints at maximum pace between the two cones/lines, with a 10-second rest in between each effort.

Main study parameters/endpoints: The primary outcome is generating reference values for the MPST for typical children aged 5-12.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: We believe the risks of experiencing drawbacks from study participation are minimal. The Muscle Power Sprint Test (MPST) is non-invasive, involving six short, consecutive 15-meter sprints - similar to activities children commonly engage in, such as games like tag or hide-and-seek - with a 10-second rest after every run. Individual testing and warm-up rounds further mitigate potential risks, and we estimate the likelihood of injuries or adverse effects to be lower than those encountered in a standard physical education class.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-12 years
* Attending primary education at one of the participating schools or attending participating after-school childcare centers.

Exclusion Criteria:

* Contra-indication for maximal exercise due to cardiac or respiratory morbidities
* Injuries limiting maximal exercise capacity
* Known with motor function impairment which may hamper maximal exercise (e.g. neurologic comorbidities)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Reference values for the MPST for children aged 5-12 years, both male and female. | Data gathering: 6 months, data processing: 6 months.
  Reference values for the MPST for children aged 5-12 years, both male and female.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Schnater, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Sophia Children's Hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
We can share the raw MPST data when requested by other researchers.

REFERENCES:
- [Background] Hijkoop A, van Schoonhoven MM, van Rosmalen J, Tibboel D, van der Cammen-van Zijp MHM, Pijnenburg MW, Cohen-Overbeek TE, Schnater JM, IJsselstijn H. Lung function, exercise tolerance, and physical growth of children with congenital lung malformations at 8 years of age. Pediatr Pulmonol. 2019 Aug;54(8):1326-1334. doi: 10.1002/ppul.24345. Epub 2019 Apr 22. PMID 31012287
- [Background] Schaan CW, Macedo ACP, Sbruzzi G, Umpierre D, Schaan BD, Pellanda LC. Functional Capacity in Congenital Heart Disease: A Systematic Review and Meta-Analysis. Arq Bras Cardiol. 2017 Oct;109(4):357-367. doi: 10.5935/abc.20170125. Epub 2017 Sep 4. PMID 28876372
- [Background] Toussaint-Duyster LCC, van der Cammen-van Zijp MHM, de Jongste JC, Tibboel D, Wijnen RMH, Gischler SJ, van Rosmalen J, IJsselstijn H. Congenital diaphragmatic hernia and exercise capacity, a longitudinal evaluation. Pediatr Pulmonol. 2019 May;54(5):628-636. doi: 10.1002/ppul.24264. Epub 2019 Feb 11. PMID 30741484
- [Background] Gischler SJ, Mazer P, Duivenvoorden HJ, van Dijk M, Bax NM, Hazebroek FW, Tibboel D. Interdisciplinary structural follow-up of surgical newborns: a prospective evaluation. J Pediatr Surg. 2009 Jul;44(7):1382-9. doi: 10.1016/j.jpedsurg.2008.12.034. PMID 19573666
- [Background] Fredriksen PM, Ingjer F, Nystad W, Thaulow E. Aerobic endurance testing of children and adolescents--a comparison of two treadmill-protocols. Scand J Med Sci Sports. 1998 Aug;8(4):203-7. doi: 10.1111/j.1600-0838.1998.tb00193.x. PMID 9764441
- [Background] Bailey RC, Olson J, Pepper SL, Porszasz J, Barstow TJ, Cooper DM. The level and tempo of children's physical activities: an observational study. Med Sci Sports Exerc. 1995 Jul;27(7):1033-41. doi: 10.1249/00005768-199507000-00012. PMID 7564970
- [Background] Stockwell S, Trott M, Tully M, Shin J, Barnett Y, Butler L, McDermott D, Schuch F, Smith L. Changes in physical activity and sedentary behaviours from before to during the COVID-19 pandemic lockdown: a systematic review. BMJ Open Sport Exerc Med. 2021 Feb 1;7(1):e000960. doi: 10.1136/bmjsem-2020-000960. eCollection 2021. PMID 34192010